CLINICAL TRIAL: NCT04167969
Title: Molecular Phenotyping and Image-Guided Surgical Treatment of Prostate Cancer Using Ultrasmall Silica Nanoparticles
Brief Title: The Use of Nanoparticles to Guide the Surgical Treatment of Prostate Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Cornell University/Weill Cornell Medical Center (Unknown); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-333
Record Dates: First submitted 2019-11-18; First posted 2019-11-19 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Prostate Cancer
Keywords: Molecular Phenotyping; Ultrasmall Silica Nanoparticles; PET/MRI; 64Cu-NOTA-PSMA-PEG-Cy5.5-C' dot tracer; (89Zr)-DFO-PSMAi-PEG-Cy5.5-C' dots; 19-333
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prostate cancer patients (Experimental): Patients will receive an intravenous (IV) injection of approximately 6-7 mCi (+/- 10%) of PSMA-targeting C' dot tracer up to 48 hours before surgery. Patients will then undergo serial preoperative PET/MR imaging to help characterize the safety, biodistribution/pharmacokinetics, and dosimetry of this agent. To assess total radioactivity in whole blood/plasma and urine samples, as well as radioactive metabolites, blood and urine samples will be collected at approximately 30 min post-injection as well as before each imaging session
  Interventions: Drug: (64Cu)-NOTA-PSMAi-PEG-Cy5.5-C' dot tracer, or (89Zr)-DFO-PSMAi-PEG-Cy5.5-C' dots; Diagnostic Test: PET/MRI/fluorescence imaging; Other: Blood and urine sampling; Procedure: laparoscopic radical prostatectomy and bilateral pelvic LN dissection or a salvage lymph node dissection

INTERVENTIONS:
Drug: (64Cu)-NOTA-PSMAi-PEG-Cy5.5-C' dot tracer, or (89Zr)-DFO-PSMAi-PEG-Cy5.5-C' dots — Patients will be injected with approximately 6-7 mCi (+/- 10%) of 64Cu-NOTA-PSMAi-PEG-Cy5.5-C' dots or 89Zr-DFO-PSMAi-PEG-Cy5.5-C' dots, up to 48 hours before surgery.
Diagnostic Test: PET/MRI/fluorescence imaging — Imaging will be performed using the GE Signa PET/MRI.
Other: Blood and urine sampling — Staff will perform the IV blood draws and collect urine samples
Procedure: laparoscopic radical prostatectomy and bilateral pelvic LN dissection or a salvage lymph node dissection — Surgery will be performed within 24 h of the third PET/MRI scan.

SUMMARY:
The purpose of this study is to see whether using the copper-64 (64Cu) or zirconium-89 (89Zr) radiolabeled PSMA-targeting C' dot tracer, termed 64Cu-NOTA-PSMAi-PEG-Cy5.5-C' dots or 89Zr-DFO-PSMAi-PEG-Cy5.5-C' dots, is a safe way to identify tumor cells before and during surgery for prostate cancer. The researchers want to determine whether pre-operative PET/MRI scans and intra-operative optical imaging performed in prostate cancer patients after the injection of one of these investigational tracers more accurately localizes cancerous deposits within the surgical bed as compared with conventional imaging scans alone. The researchers will study how the tracer travels through your body and where it is distributed. This study is the first time that the tracer will be used in patients undergoing surgery for prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

Primary RP + PLND

* Age ≥18 years
* Patients meeting one of the following criteria:

  * Tumor clinical stage T3a or higher
  * Gleason score 8-10, or
  * PSA level > 20 ng/mL
* Patients deemed fit for surgery on the basis of preoperative evaluation at the physician's discretion
* Patient is scheduled for standard of care laparoscopic radical prostatectomy (with or without robotic assistance)

Salvage PLND

* Age ≥18 years
* Patients with presence of suspicious lymph node on CT or MRI (of a pelvic node => 10mm in short axis or a node with abnormal morphology such as roundness irregularity or loss of fatty hilum, or PSMA-avid on PSMA PET imaging
* Patients deemed fit for surgery on the basis of preoperative evaluation at the physician's discretion
* Patient is scheduled for standard of care salvage pelvic lymph node dissection (with or without robotic assistance)

Exclusion Criteria:

* Contraindications to standard-of-care MR imaging (e.g., metal implants, claustrophobia)
* Prior androgen-deprivation therapy for prostate cancer (N/A for Salvage PLND)
* Prior pelvic radiotherapy (N/A for Salvage PLND )
* Medical illness unrelated to the tumor that, in the opinion of the attending physician and principal investigator, will preclude administration of the tracer

  °This includes patients with uncontrolled infection, chronic renal insufficiency (EGFR < 60 mL/min/1.73m2), myocardial infarction within the past 6 months, unstable angina, cardiac arrhythmias other than chronic atrial fibrillation and chronic active or persistent hepatitis, or New York Heart Association Classification III or IV heart disease
* Weight greater than the 400-lb weight limit of the PET scanner
* Unmanageable claustrophobia
* Inability to lie in the scanner for 30 min

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer
Enrollment: 16 (Estimated)
Dates: Start 2021-02-17 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Side effects | 1 year
  Will be described using CTCAE version 5 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Karim Touijer, MD, MPH, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm